CLINICAL TRIAL: NCT02664987
Title: A Cross-sectional Study to Investigate the Pain Control Status in Cancer Patients in South East Asian Countries
Brief Title: Analgesic Treatment for Cancer Pain in South East Asia
Acronym: ACE
Status: Completed | Type: Observational
Sponsor: Mundipharma Pte Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: OPD14-AP-401
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: Pain
Keywords: pain management, pain control, cancer
MeSH Terms: conditions — Pain; Agnosia; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving cancer pain treatment
  Interventions: Other: Patients receiving cancer pain treatment

INTERVENTIONS:
Other: Patients receiving cancer pain treatment

SUMMARY:
This study is planned to investigate the pain control status in cancer patients in 6 South East Asian countries through evaluation of prescription pattern of analgesics, satisfaction of pain control, quality of life and assessment of the adequacy of pain control and relationship among these factors in cancer patients with pain. Cancer pain is undermanaged and it is hoped that this study will be used as a reference for effective cancer pain management in these countries.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (over 18 years) cancer patients [country variation would be accepted based on the definition of adults]
2. Cancer has been diagnosed pathologically
3. Out-patients with cancer pain due to cancer itself or its treatment
4. Patients being treated with any analgesics for more than one month for the management of cancer pain at enrolment
5. Patients who are willing to voluntarily sign the study consent form

Exclusion Criteria:

1. Patients who have had an operation for any reasons within 3 months prior to the enrolment
2. Patients with any oncologic emergency
3. Patients who had any interventional therapy (e.g. nerve block, neurolytic procedures) related to their cancer pain within 6 weeks of study entry
4. Insufficient ability or willingness to cooperate
5. Patients who are judged not suitable to participate in this study by the investigator
6. Patients who are participating in any other interventional clinical trials for cancer treatment or supportive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects were selected from government and private hospitals that see cancer patients.
Sampling Method: Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

REFERENCES:
- [Derived] Thinh DHQ, Sriraj W, Mansor M, Tan KH, Irawan C, Kurnianda J, Nguyen YP, Ong-Cornel A, Hadjiat Y, Moon H, Javier FO. Analgesic Prescription Patterns and Pain Outcomes in Southeast Asia: Findings From the Analgesic Treatment of Cancer Pain in Southeast Asia Study. J Glob Oncol. 2018 Sep;4:1-10. doi: 10.1200/JGO.17.00055. PMID 30241271
- [Derived] Thinh DHQ, Sriraj W, Mansor M, Tan KH, Irawan C, Kurnianda J, Nguyen YP, Ong-Cornel A, Hadjiat Y, Moon H, Javier FO. Patient and Physician Satisfaction with Analgesic Treatment: Findings from the Analgesic Treatment for Cancer Pain in Southeast Asia (ACE) Study. Pain Res Manag. 2018 Apr 18;2018:2193710. doi: 10.1155/2018/2193710. eCollection 2018. PMID 29849841

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Receiving Cancer Pain Treatment: Single arm -- Patients receiving cancer pain treatment
Period: Overall Study
Arm/Group | Patients Receiving Cancer Pain Treatment
Started | 462
Completed | 462
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Receiving Cancer Pain Treatment
Number analyzed (Participants) | 462
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.14 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248
  Male | 214

OUTCOME MEASURES:

1. Primary Outcome: Prescription Pattern of Analgesics (Opioid or Non-opioid)
Description: At Visit 1 (Day 1) which was the only visit in the study, data was collected on whether each patient was receiving only opioid, only non-opioid or both opioid and non-opioid analgesic treatments for pain control.
Time Frame: Day 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Patients Receiving Cancer Pain Treatment
Number analyzed (Participants) | 462
percentage of patients
  Opioid analgesics only | 37.27 [31.83 to 42.92]
  Non-opioid analgesics only | 11.33 [7.58 to 15.31]
  Opioid and non-opioid analgesics | 51.40 [46.13 to 56.83]

2. Primary Outcome: Satisfaction With Patient's Pain Control as Measured by 5-point Scale Answered by Patients and Investigators
Description: The scale used to measure a patient's satisfaction with pain control ranges from 1 to 5:
  1. Very satisfied
  2. Satisfied
  3. Acceptable
  4. Dissatisfied
  5. Very dissatisfied
  Patients and Investigators will each indicate their opinion on separate scales.
Time Frame: Day 1
Measure: Number; unit: percentage of patients
Arm/Group | Patients Receiving Cancer Pain Treatment
Number analyzed (Participants) | 462
percentage of patients
  Very satisfied- answered by patient | 18.6
  Satisfied- answered by patient | 41.6
  Acceptable- answered by patient | 30.3
  Dissatisfied- answered by patient | 8.0
  Very dissatisfied- answered by patient | 1.5
  Very satisfied- answered by Investigator | 12.1
  Satisfied- answered by Investigator | 42.0
  Acceptable- answered by Investigator | 25.3
  Dissatisfied- answered by Investigator | 19.1
  Very dissatisfied- answered by Investigator | 1.5

3. Primary Outcome: Quality of Life as Measured Using EQ-5D-3L Questionnaire Answered by Patient
Description: EQ-5D-3L summary indices were calculated using the algorithm developed based on the valuation of EQ-5D-3L health states from an adult Thai population (Tongsiri & Cairns, 2011). Applying the Thai algorithm, EQ-5D-3L summary indices range from -0.45 to 0.80, with an EQ-5D-3L summary index of 0.80 indicating the best overall health-related quality of life.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Receiving Cancer Pain Treatment
Number analyzed (Participants) | 462
units on a scale | 0.45 (0.30)

4. Primary Outcome: Intensity of Pain Currently and Over Past 24 Hours as Measured by NRS Scores Indicated by Patient
Description: Patients indicated their pain intensity using a numerical rating scale (NRS) ranging from 0 (no pain) to 10 (worst possible pain).
  Their current pain intensity and pain in the last 24 hours were indicated on separate scales. A higher score indicates higher pain intensity.
Time Frame: Past 1 day up to Day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Receiving Cancer Pain Treatment
Number analyzed (Participants) | 462
units on a scale
  Current pain intensity level | 4.10 (2.61)
  Pain intensity level in the last 24 hours | 4.76 (2.47)

5. Secondary Outcome: Sleep Disturbance Within Last 7 Days Assessed Using Questionnaire Answered by Patient
Description: Patients answered "yes" or "no" to the following question:
  "Have you had trouble sleeping due to your cancer pain within the last 7 days?"
Time Frame: Past 7 days up to Day 1
Measure: Number; unit: percentage of patients
Arm/Group | Patients Receiving Cancer Pain Treatment
Number analyzed (Participants) | 462
percentage of patients
  No trouble sleeping | 45.2
  Had trouble sleeping | 54.8

6. Secondary Outcome: Patient's Performance Status as Measured by Investigator's Rating on ECOG PS Scale
Description: The Eastern Cooperative Oncology Group Performance Status (ECOG PS) scale ranges from 0 to 4:
  0- Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  A higher score indicates greater functional impairment.
Time Frame: Day 1
Measure: Number; unit: percentage of patients
Arm/Group | Patients Receiving Cancer Pain Treatment
Number analyzed (Participants) | 462
percentage of patients
  0- Fully active | 14.9
  1- Restricted strenuous activity | 42.7
  2- Ambulatory | 26.6
  3- Limited self-care | 13.6
  4- Completely disabled | 2.2

ADVERSE EVENTS:
Description: This is an observational study with no investigational product involved. Therefore, there were no serious and non-serious adverse events collected and assessed as part of the study.
Arm/Group | Patients Receiving Cancer Pain Treatment
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator may not publish the results of the study without prior approval from Mundipharma.